CLINICAL TRIAL: NCT07402785
Title: The Effect of Abdominal Massage on Constipation in Patients Receiving Hemodialysis Treatment
Brief Title: The Effect of Abdominal Massage on Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat Tukenmez (Other)
Responsible Party: Sponsor-Investigator, Firat Tukenmez, NURSE, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTU-SBE-FT-01
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hemodialysis; Constipation
Keywords: abdominal massage
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled clinical trial with an experimental, pretest-posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (n = 25) (No Intervention): The control group did not receive abdominal massage and continued their routine treatment. In groups, outcome measures were assessed at baseline (first week) and at the end of the study period (sixth week). For evaluation Bristol Stool Form Scale, Constipation Severity Scale, and Constipation Quality of Life Questionnaire, administered face-to-face by the researcher.
- intervention group (n = 24) (Experimental): One patient in the intervention group died one month after the initiation of the study, and the intervention was discontinued for this patient.Abdominal massage was administered to the intervention group during hemodialysis sessions in the dialysis units of the respective hospitals, without interrupting the treatment process. Patient privacy was ensured using a curtain before each session. Massage was applied at least 30 minutes after meals. Before each session, patients' general physical and mental condition, vital signs, abdominal tension/sensitivity, and skin integrity were assessed.
  Abdominal massage was performed by the researcher twice weekly for six weeks, with each session lasting 15 minutes, for a total of 12 sessions. At the end of the sixth week, the effectiveness of the intervention was evaluated using the Bristol Stool Form Scale, Constipation Severity Scale, and Constipation Quality of Life Questionnaire, administered face-to-face by the researcher.
  Interventions: Other: abdominal massage

INTERVENTIONS:
Other: abdominal massage — Abdominal massage is considered a promising complementary approach for alleviating the symptoms of chronic constipation due to its noninvasive nature and relatively low cost. This intervention is thought to stimulate somato-autonomic reflexes and intestinal motility, thereby enhancing peristalsis and promoting contractions of the rectal muscles. Through massage application, bowel movements become more active. In addition, abdominal massage exerts effects on the abdominal muscles and the large intestine, and by stimulating the abdominal nerve plexus (splanchnic plexus), it alters intestinal tone. As a result of these mechanisms, constipation-related symptoms such as pain and discomfort are reduced.
  Arms: intervention group (n = 24)

SUMMARY:
This study aimed to determine the effect of abdominal massage on constipation in patients undergoing hemodialysis. The main questions he intends to answer are:

H0: Abdominal massage applied to patients undergoing hemodialysis treatment has no effect on constipation. H1: Abdominal massage applied to patients receiving hemodialysis treatment has an effect on constipation.

DETAILED DESCRIPTION:
Participants and Setting The study population consisted of patients receiving hemodialysis treatment at the Dialysis Units of Rize Training and Research Hospital and Rize State Hospital. A total of 50 patients who met the inclusion criteria and did not meet any exclusion criteria were included in the study.

Eligible patients (n = 50) were listed and randomly assigned to either the intervention group (n = 25) or the control group (n = 25) using a simple randomization method via a computer-based program (https://randomizer.org/). One patient in the intervention group died one month after the initiation of the study, and the intervention was discontinued for this patient. Consequently, the study was completed with 49 patients (intervention group, n = 24; control group, n = 25).

Intervention and Control Prior to the study, the researcher completed a structured training program consisting of 16 hours of theoretical education and 24 hours of practical training provided by the Department of Physical Therapy and Rehabilitation at Rize Training and Research Hospital. An official certificate confirming completion of this training was issued by the hospital administration.

Abdominal massage was administered to the intervention group during hemodialysis sessions in the dialysis units of the respective hospitals, without interrupting the treatment process. Patient privacy was ensured using a curtain before each session. Massage was applied at least 30 minutes after meals. Before each session, patients' general physical and mental condition, vital signs, abdominal tension/sensitivity, and skin integrity were assessed.

Abdominal massage was performed by the researcher twice weekly for six weeks, with each session lasting 15 minutes, for a total of 12 sessions. At the end of the sixth week, the effectiveness of the intervention was evaluated using the Bristol Stool Form Scale, Constipation Severity Scale, and Constipation Quality of Life Questionnaire, administered face-to-face by the researcher.

The control group did not receive abdominal massage and continued their routine treatment. In both groups, outcome measures were assessed at baseline (first week) and at the end of the study period (sixth week).

Statistical Analysis Data were analyzed using the Statistical Package for the Social Sciences (SPSS) for Windows, version 26.0. Distribution characteristics were assessed using skewness and kurtosis values, all of which ranged between -2 and +2, indicating normal distribution. Descriptive statistics (frequency, percentage, mean, median, and standard deviation) were used. Independent t-tests were employed for between-group comparisons, paired t-tests for within-group comparisons, and the chi-square test for categorical variables. Parametric statistical methods were applied, and a p-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Voluntarily agreed to participate in the study
* Receiving hemodialysis treatment for at least one month
* Diagnosed with constipation by a clinician or meeting Rome IV criteria
* Able to communicate effectively and respond to all study-related questions, either personally or through a caregiver

Exclusion Criteria:

* History of ileus or intestinal perforation
* Presence of abdominal distension
* Presence of a colostomy or ileostomy
* Presence of extensive abdominal skin disease or infection
* Diagnosis of inflammatory bowel disease
* Presence of signs or symptoms of an acute abdomen
* Presence of diarrhea
* Known allergy to baby oil
* Refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-08-09 (Actual)

PRIMARY OUTCOMES:
Constipation Severity | baseline and end of week 6
  change in constipation severity measured using the Constipation Severity Scale

SECONDARY OUTCOMES:
Constipation-related Quality of Life | Baseline and end of week 6
  Change in quality of life measured using the Constipation Quality of Lise Questionnaire.
Stool Consistency | Baseline and end of week 6
  Stool from assessed using the Bristol Stool Form Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Confidentiality of the study Participant confidentiality was strictly maintained throughout the study. All personal and clinical data were anonymized by assigning unique identification codes to each participant, and no identifying information was included in the data collection forms or analysis. Study data were accessible only to the research team and were stored securely in accordance with institutional and ethical guidelines. The results were reported in aggregate form to ensure that individual participants could not be identified.

REFERENCES:
- See also: Related Info — https://www.nih.gov